CLINICAL TRIAL: NCT06297824
Title: Can a Brief Emotion Regulation Group Therapy Help Adolescents With Deliberate Self-Harm? A Feasibility Study and a Qualitative Interview Study
Brief Title: Feasibility of Emotion Regulation Group Therapy for Adolescent Self-Harm
Acronym: ERGT-A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Hanna Sahlin, Principal Investigator, PhD, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-04909-01
Record Dates: First submitted 2024-01-29; First posted 2024-03-07 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Self-harm; Emotion Regulation; Adolescent - Emotional Problem
Keywords: self-harm; Emotion regulation; Group treatment; Adolescents
MeSH Terms: conditions — Self-Injurious Behavior; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: Feasibility, open trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ERGT-A (Other): 12 session emotion regulation treatment in group format. Psychoeducation and homework assignments. Subjects taught are the function of deliberate self-harm (DSH), functionality of emotions, negative consequences of emotional avoidance, non-avoidant emotion regulation.
  Interventions: Behavioral: ERGT-A

INTERVENTIONS:
Behavioral: ERGT-A — Emotion regulation group therapy for adolescents

SUMMARY:
Deliberate self-harm (DSH) is a prevalent behaviour among adolescents but there is no current recommendation for an efficacious treatment. Emotion regulation group therapy (ERGT) is a brief treatment for DSH with a well-documented utility and feasibility in the adult population, and an adapted version for adolescents may provide equal benefits for adolescents, provided adjustments to prevent or decrease social contagion are present.

A quantitative feasibility open trial (N=20) followed up by a qualitative interview study will examine the feasibility, acceptability and preliminary effect of ERGT for adolescents.

DETAILED DESCRIPTION:
Deliberate self-harm (DSH) is a prevalent behaviour among adolescents but there is no current recommendation for an efficacious treatment. Emotion regulation group therapy (ERGT) is a brief treatment for DSH with a well-documented utility and feasibility in the adult population, and an adapted version for adolescents may provide equal benefits for adolescents, provided adjustments to prevent or decrease social contagion are present. Adaptations to ERGT will result in a 12 session long treatment for adolescents Emotion regulation group therapy for Adolescents (ERGT-A). A parallel parent group focused on strengthening parental skills will be given alongside ERGT-A (5 sessions)

Method: A quantitative feasibility open trial (N=20) with pre, post and 1 month follow-up assessments will examine the feasibility, acceptability and preliminary effect of ERGT for adolescents.

Feasibility measures include recruitment rate, proportion beginning treatment, attrition, treatment credibility and satisfaction, negative effects, and alliance.

Preliminary effects measures include DSH, emotion regulation ability, anxiety and depression.

Method: A qualitative interview study. Using thematic analysis to explore participants' experience of ERGT-A and parent group

ELIGIBILITY:
Inclusion Criteria:

1. 13-17 years of age;
2. having engaged in deliberate self-harm (DSH)-behaviours ≥ 5 times the last year;
3. having engaged in ≥1 DSH episode during the past month;
4. having ongoing psychiatric treatment in the community;
5. having at least one caregiver or other significant adult, committed to participate in the parent program; and
6. stability of psychotropic medications

Exclusion Criteria:

1. a diagnosis of psychotic, bipolar I disorder or severe social anxiety disorder (SAD);
2. ongoing substance dependence;
3. the presence of co-occurring psychiatric disorders that require immediate treatment;
4. having an autism spectrum disorder together with borderline intellectual disability or having an intellectual disability;
5. insufficient understanding of the Swedish language

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
Feasibility measure, recruitment rate | through study completion, an average of 1 year
  Recruitment rate
Feasibility measures, proportion included | through study completion, an average of 1 year
  Proportion of participants invited to participate who accepts and is included (higher = better, min 0%- max 100%)
Feasibility measures, compliance | Pre-treatment to post-treatment (End of treatment, EOT) (12 weeks)
  Compliance, no of sessions attended (>50%), (higher = better, min 0-max 10)
Feasibility measures, attrition | Pre-treatment to post-treatment EOT (12 weeks)
  Attrition, percent of included participants who drops out of treatment (lower = better, min 0%- max 100%)
Feasibility measures, client satisfaction | at post-treatment EOT (12 weeks)
  Mean score on Client satisfaction questionnaire> 25 (higher= better, min 8-max 32)
Feasibility measures, negative effects of treatment | at post-treatment EOT (12 weeks)
  Low rating on Negative effects Questionnaire (lower= better, min 0-max 20)

SECONDARY OUTCOMES:
Preliminary effect, self harm frequency EOT | Pre-treatment to post-treatment (EOT) (12 weeks)
  Mean Deliberate self-harm frequency at post-treatment (min 0-max 100, lower=better)
Preliminary effect, self harm frequency 1MFU | Post-treatment (EOT) to follow-up (4 weeks)
  Mean Deliberate self-harm frequency at post-treatment and 1MFU lower than at post-treatment (min 0-max 100, lower=better)
Preliminary effect, emotion dysregulation EOT | Pre-treatment to post-treatment (EOT) (12 weeks)
  Mean difficulty in emotion regulation rating (DERS-16) at post-treatment lower than at pre-treatment (min 16, max 80, lower=better)
Preliminary effect, emotion dysregulation 1MFU | Post-treatment (EOT) to follow-up (4 weeks)
  Mean difficulty in emotion regulation rating (DERS-16) at 1MFU lower than at post-treatment (min 16, max 80, lower=better)

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Sahlin, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Prima Barn och Vuxenpsykiatri Handen och Järva, Stockholm, Spånga, Sweden

IPD SHARING:
Plan to Share IPD: No